CLINICAL TRIAL: NCT07167680
Title: Development and Validation of a mHealth Fall Management Program - Phase III
Brief Title: Fall Prevention Among People With Spinal Cord Injury and Multiple Sclerosis Who Use Wheelchairs and Scooters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Laura Rice, Associate Professor in the Department of Health and Kinesiology; Associate Head for Graduate Studies; Associate Director of the Center for Health, Aging, and Disability; Principal Investigator, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB25-0827; 90DPHF0010 (Other Grant/Funding Number: NIDILRR); 862958 (Other Grant/Funding Number: Craig H. Neilsen Foundation)
Record Dates: First submitted 2025-08-08; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries (SCI); Multiple Sclerosis
Keywords: wheelchair; fall prevention; mobile application; spinal cord injury; multiple sclerosis; education
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis | interventions — Death Domain

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two arms in a parallel design: (1) Fall prevention education via the iROLL program or (2) Fall prevention education via the STEADI program. Each participant remains in their assigned group throughout the study.
Who Masked: Participant
Masking Description: Participants will be blindly assigned to one of the groups to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized reduction of falls (iROLL) Group (Experimental): iROLL group participants will be educated about fall prevention and management strategies using the individualized reduction of falls (iROLL) mobile application (app)
  Interventions: Procedure: Individualized reduction of falls (iROLL)
- Stopping Elderly Accidents, Deaths & Injuries (STEADI) Program Group (Active Comparator): STEADI group participants will be educated about fall prevention and management strategies using Centers for Disease Control and Prevention entitled: Stopping Elderly Accidents, Deaths & Injuries (STEADI) program.
  Interventions: Procedure: Stopping Elderly Accidents, Deaths & Injuries (STEADI)

INTERVENTIONS:
Procedure: Individualized reduction of falls (iROLL) — The iROLL program is a 6-week fall prevention and management program for people living with spinal cord injury (SCI) and multiple sclerosis (MS) who use wheelchairs and scooters. The program's overall goals are to reduce fall frequency, improve functional mobility skills, decrease fear of falling, increase quality of life, and increase community participation. It uses many active learning strategies such as: goal setting, journaling, small group discussions, practicing skills, and homework to apply content to one's daily life.
  Arms: Individualized reduction of falls (iROLL) Group
Procedure: Stopping Elderly Accidents, Deaths & Injuries (STEADI) — The CDC's Stopping Elderly Accidents, Deaths & Injuries (STEADI) initiative is a coordinated approach to fall prevention for older adults. It focuses on helping healthcare providers implement clinical fall prevention strategies, including screening for fall risk, assessing modifiable risk factors, and intervening to reduce risk.
  Arms: Stopping Elderly Accidents, Deaths & Injuries (STEADI) Program Group

SUMMARY:
The research team is conducting a study to determine if a fall prevention program designed specifically for people who use wheelchairs and scooters can help people better prevent and manage falls compared to the standard of care.

This study will compare two groups of participants:

1. One group will use the iROLL-O+ app, which offers personalized fall prevention tools and strategies.
2. The other group will receive fall prevention information from a well-known program developed by the Centers for Disease Control and Prevention (CDC), called STEADI, which stands for Stopping Elderly Accidents, Deaths, and Injuries.

This study includes adults living with Spinal Cord Injury (SCI) or Multiple Sclerosis (MS) who use a wheelchair or scooter every day. The research team aims to determine which approach is more effective in reducing falls and improving confidence in performing daily activities.

DETAILED DESCRIPTION:
People living with SCI or MS who use wheelchairs and scooters (WC/S) full time often experience falls. In fact, 7 out of 10 report falling at least once every 6 to 12 months. These falls can lead to serious injuries and emotional distress, such as concerns about falling (CaF). Although falls are common among this population, most fall prevention programs are designed for people who can walk. There are very few programs designed for people who use WC/S.

This study will test to see if a fall prevention and management program designed specifically for people who use WC/S does a better job at helping people learn how to prevent and manage falls compared to a program that is designed for older adults.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older.
* History of Multiple Sclerosis (MS) or Spinal Cord Injury (SCI).
* Able to transfer independently or with minimal to moderate assistance.
* Unable to walk 25 feet or more
* Have experienced at least 1 fall in the past three years.
* Have a care partner to assist the participant when practicing physical skills.
* Have access to a smartphone/iPad.
* Have a stable internet connection.

Exclusion Criteria:

* Multiple sclerosis exacerbation in the past 30 days, or are unable to remain in an upright position for an hour.
* Impaired cognition (a score of 10 or above on the Short Blessed Test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Currently Employed Technology Scale | Baseline
  Assesses how individuals with disabilities utilize currently available and assistive technologies in their everyday lives across five functional domains (Home, Social, E-commerce, Health Care, Technical).
  Subscale (Domain)
  Scoring:
  Each domain's subtotal ranges from 0 to 10. Higher scores indicate more frequent use of technology.
  Interpretation categories:
  0-2: Very Infrequent IT Use; 3-4: Infrequent IT Use; 5-6: Moderate IT Use; 7-8: Frequent IT Use; 9-10: Very Frequent IT Use
  Total FACETS Score:
  Ranges from 0 to 50 (sum of the five domain subtotals). Higher total scores = greater overall frequency of technology use.
  Interpretation categories:
  0-14: Very Infrequent IT Use; 15-24: Infrequent IT Use; 25-34: Moderate IT Use; 35-44: Frequent IT Use; 45-50: Very Frequent IT Use
Fall Concerns Scale for Wheelchair and Scooter Users | Baseline, Post-Intervention (Week 6 and Week 14)
  Measures fear of falling and fall-related self-efficacy in individuals who use wheelchairs or scooters. The Fall Concerns Scale for Wheelchair and Scooter Users consists of 16 items, each rated on a 4-point Likert scale (1 = "not at all concerned" to 4 = "very concerned"). The total score ranges from 16 to 64, with higher scores indicating greater fear of falling and lower fall-related self-efficacy.
Falls Prevention Strategies Survey | Baseline, Post-Intervention (Week 6 and Week 14)
  Captures the frequency and types of fall prevention behaviors or strategies participants use in their daily lives.
The Fall Management Scale | Baseline, Post-Intervention (Week 6 and Week 14)
  Assesses participant confidence and preparedness in managing fall-related scenarios (e.g., recovery techniques, communication, and safety). Total scores range from 0 to 64. Higher scores indicate greater use of fall management strategies (better outcome).
Fall Prevention and Management Questionnaire | Baseline, Post-Intervention (Week 6 and Week 14)
  A multi-dimensional tool that evaluates participants' knowledge, behaviors, and attitudes toward fall prevention and recovery.
Community Participation Indicators Questionnaire | Baseline, Post-Intervention (Week 6 and Week 14)
  A self-report 48-item objective that measures two distinct subsets:
  1) Importance and meaning, and 2) Control over participation. This questionnaire assesses levels of community engagement, social interaction, and participation in everyday activities outside the home. Items are typically rated on a Likert scale and aggregated to produce subscale scores and a total participation score.
  Higher scores indicate greater community participation.
  Scores range between 0 and 1, where:
  0 = no meaningful participation.
  1 = full participation in all important activities
Transfer Assessment Instrument Questionnaire | Baseline, Post-Intervention (Week 6 and Week 14)
  Measures participants' safety, technique, and confidence when transferring between surfaces (e.g., wheelchair to bed).
Wheelchair Skills Test - Questionnaire | Baseline, Post-Intervention (Week 6 and Week 14)
  Self-reported version of the Wheelchair Skills Test assessing wheelchair handling and maneuvering capabilities.
System Usability Scale | Post-Intervention (Week 6)
  Evaluates participants' perceived usability of the iROLL-O+ mobile app - only for the intervention group.
  The SUS consists of 10 items, each scored on a 5-point Likert scale (0-4). The total raw score is converted to a 0-100 scale.
  Higher scores indicate better usability. A score of 68 is considered average usability; scores above 68 reflect above-average usability, while scores below 68 reflect below-average usability.
Usefulness, Satisfaction, and Ease of Use Questionnaire | Post-Intervention (Week 6)
  Assesses perceived usefulness, satisfaction, and ease of use of a mobile app. - only for the intervention group
Mobile App Rating Scale | Post-Intervention (Week 6)
  Evaluates mobile app quality, including engagement, functionality, aesthetics, and information content. - Only for the intervention group.
  The uMARS contains 20 items across four objective quality subscales (Engagement, Functionality, Aesthetics, Information).
  Each item is rated on a 5-point Likert scale (1-5). Subscale scores are averaged, and a total quality mean score can also be calculated.
  Higher scores indicate higher app quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Disability Participation and Quality of Life (DPQOL) Laboratory, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, an IRB-approved research team member (research assistant) will create a copy of the original data. All the identifiable information will be redacted from both online surveys and interview transcripts and unique codes will be assigned to each participant data. The identifiable data will be saved separately in a secure UIUC Box folder and only the de-identified data will be submitted to a data repository (Inter-university Consortium for Political and Social Research - ICPSR).
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Start date: after completion of the study; End date: NA
Access Criteria: The data will be retrieved through the ICPSR platform, which provides secure access to the research datasets. Access is limited to individuals affiliated with ICPSR member institutions or those who obtain direct permission/licensing through ICPSR.
URL: https://www.icpsr.umich.edu/sites/icpsr/manage-data